CLINICAL TRIAL: NCT01619566
Title: Duloxetine (Cymbalta): for Fibromyalgia: An Open Label Study to Assess Potential Mechanisms for Fibromyalgia in Peripheral Tissue Innervation That Could Predict Therpeutic Responsiveness to Duloxetine.
Brief Title: Cymbalta for Fibromyalgia Pain - Predictive Value of Small Fiber Changed
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor related
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Tobias Moeller-Bertram, Associate Clinical Professor of Anesthesia, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111654
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Duloxetine; Cymbalta; Pain; Peripheral Nerve; Biopsy; Predictive
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Control subjects undergo a skin biopsy.
- Treatment (Experimental): Subjects in the treatment arm also undergo a skin biopsy, followed by 8 week treatment with Duloxetine.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — oral tablet, 30mg daily for 1 week (titration up) oral tablet, 60mg daily for 8 weeks (treatment) oral tablet, 30mg daily for 1 week (titration down, if needed)
  Other Names: Cymbalta
  Arms: Treatment

SUMMARY:
Subjects with Fibromyalgia who respond to Duloxetine have specific nerve fiber characteristics. This can be used to predict which future patients will respond to Duloxetine.

DETAILED DESCRIPTION:
Subjects will have skin biopsies taken and evaluated for specific pathologies. All subjects will undergo a treatment period with Duloxetine. The analysis will correlate treatment effectiveness with pathological skin biopsy findings to predict future treatment success.

ELIGIBILITY:
Inclusion Criteria: Treatment Arm

* Fibromyalgia Diagnosis
* Female
* Over the age of 18, under the age of 70
* Understands English
* Not Pregnant/planning to become pregnant

Exclusion Criteria:

* No major psychiatric disorders
* No major unconrolled systemic diseases which may require hospitalization in the next 6 months
* Pregnant

Inclusion Criteria: Control Arm

* Female
* Over the age of 18, under the age of 70
* Understands English
* Not Pregnant/planning to become pregnant

Exclusion Criteria: Control Arm

* No major psychiatric disorders
* No major unconrolled systemic diseases which may require hospitalization in the next 6 months
* Pregnant

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Pain Reduction | 12 weeks
  Changes in Pain measured by Numeric Pain Rating Scale over time. The Numeric Pain Rating Scale (NPRS) is assessing the patients pain on a 11-point rating scale from 0 - 10 with 0 being no pain at all and 10 being the worst imaginable pain. The test is self-reported and can also be administered by an interviewer.

CONTACTS AND LOCATIONS:
Overall Officials: tobias moeller-bertram, MD, Principal Investigator — employee
Locations (1):
- University of California, San Diego Medical Centers, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Drug manufacturers website for study drug — http://www.cymbalta.com/Pages/index.aspx
- See also: Website for location of study — http://health.ucsd.edu